CLINICAL TRIAL: NCT02977598
Title: Association Between Atherogenic Index of Plasma, Blood Pressure and Impaired Glucose Metabolism
Brief Title: Relations Between Atherogenic Index of Plasma-Glucose Metabolism
Status: Completed | Type: Observational
Sponsor: Erzincan University (Other)
Responsible Party: Principal Investigator, HILAL ALPCAN, Internal medicine, medical doctor, Erzincan University
Other Study IDs: 44495147/1-202
Record Dates: First submitted 2016-11-20; First posted 2016-11-30 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus Risk

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- non-diabetic: According to the 75 g oral glucose tolerance test participants were categorized into the three groups; non-diabetic, prediabetic, and diabetic based on the criteria of the American Diabetes Association.
- prediabetic: According to the 75 g oral glucose tolerance test participants were categorized into the three groups; non-diabetic, prediabetic, and diabetic based on the criteria of the American Diabetes Association.
- diabetic: According to the 75 g oral glucose tolerance test participants were categorized into the three groups; non-diabetic, prediabetic, and diabetic based on the criteria of the American Diabetes Association.

SUMMARY:
In this study, the investigators aimed to find out whether there is any association between the atherogenic index of plasma with the glucose metabolism.In this respect, apart from the well-known diabetic risk factors, the investigators purposed to reveal new ones.

DETAILED DESCRIPTION:
Atherogenic index of plasma (AIP) is a relatively new index and a predictor of cardiovascular risk. AIP has been shown to be associated with impaired glucose metabolism. This study aimed to evaluate the relationship between AIP and parameters of glucose metabolism.

Methods: This observational study involved 448 healthy individuals who were at risk for diabetes. They were sent to hospital for diabetes check. According to the 75 g oral glucose tolerance test participants were categorized into the three groups; non-diabetic, prediabetic, and diabetic based on the criteria of the American Diabetes Association (ADA). The association between the diabetes group, AIP and parameters of glucose metabolism was analyzed.

The accuracy of registry data compatible with medical records. Statistical analyses were carried out using the Statistical Package for Social Sciences, Windows version 15.0 (SPSS, Chicago, Illinois, USA). Descriptive statistics for each variable were determined. Normality of the data distribution was assessed with the Kolmogorov-Smirnov test. For continuous variables, non-parametric statistics (Mann-Whitney or Kruskal-Wallis), and parametric statistics (t-test, ANOVA analysis) were used as appropriate. Statistically significant differences between the groups were determined by the chi-square test for categorical variables. Associations between the variables were explored using the Pearson correlation and Spearman's rho (for data that was not normally distributed). Linear regression analysis with backward elimination was also performed to define variables associated with AIP.

ELIGIBILITY:
Inclusion Criteria:

* All the participants were previously healthy, aged between 18 and 80 years, and were at risk for diabetes according to new criteria provided by the American Diabetes Association.

Exclusion Criteria:

* Individuals with a history of chronic medical diseases and those who reported current use of any medication were excluded from the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 448 healthy individuals who were at risk for diabetes. According to the 75 g oral glucose tolerance test participants were categorized into the three groups; non-diabetic, prediabetic, and diabetic based on the criteria of the American Diabetes Association.
Sampling Method: Non-Probability Sample
Enrollment: 448 (Actual)
Dates: Start 2014-02; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Atherogenic index of plasma (AIP) values compared with glucose metabolism parameters like HbA1c, Fasting Plasma Glucose and 2-hour plasma glucose levels. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: EMIN MURAT AKBAS, Assoc. Prof., Principal Investigator — ERZINCAN MENGUCEKGAZI TRAINING AND RESEARCH HOSPİTAL DEPARTMENT OF ENDOCRINOLOGY AND METABOLIC DISEASES
Locations (2):
- Turkey (Türkiye) (2):
  - Erzincan Mengucekgazi Research and Training Hospital, Erzincan
  - Erzincan Mengücekgazi Training and Research Hospital, Erzincan

IPD SHARING:
Plan to Share IPD: No